CLINICAL TRIAL: NCT01612507
Title: A Phase I, Single Centre, Randomised, Double-blind, Placebo-controlled Parallel Group Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ceftaroline After Different Intravenous Dose Regimens of Ceftaroline Fosamil to Healthy Subjects
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of Ceftaroline in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3720C00010
Record Dates: First submitted 2012-06-04; First posted 2012-06-05 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; healthy volunteers; Parallel Group Study; ceftaroline fosamil different doses; safety; Cmax; tmax; AUC
MeSH Terms: interventions — Ceftaroline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- A (Experimental): 600 mg Ceftaroline fosamil 1 h infusion
  Interventions: Drug: 600 mg Ceftaroline fosamil
- B (Experimental): Placebo 1 h infusion
  Interventions: Drug: Placebo
- C (Experimental): 600 mg Ceftaroline fosamil 2 h infusion
  Interventions: Drug: 600 mg Ceftaroline fosamil
- D (Experimental): Placebo 2 h infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 600 mg Ceftaroline fosamil — 1 h infusion
  Arms: A
Drug: Placebo — 1 h infusion
  Arms: B
Drug: 600 mg Ceftaroline fosamil — 2 h infusion
  Arms: C
Drug: Placebo — 2 h infusion
  Arms: D

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of different dose regimens of Ceftaroline

DETAILED DESCRIPTION:
A Phase I, Single Centre, Randomised, Double-blind, Placebo-controlled Parallel Group Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ceftaroline after Different Intravenous Dose Regimens of Ceftaroline Fosamil to Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures including the optional safety biomarker analysis
* Healthy male and female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture
* Women of childbearing potential must have a negative pregnancy test, be non-lactating, and be using a highly effective form of birth control for 1 month prior to enrollment, during the study, and for 3 months after completion of all study-related proceed
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg

Exclusion Criteria:

* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 3 months of the first administration of investigational drug
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV)
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant abnormalities in the physical examination, 12-lead ECG, or vital signs, as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in terms of adverse events, laboratory data, vital signs following single and multiple dose regimens of ceftaroline fosamil compared to placebo | Screening up to 19 days after first dose

SECONDARY OUTCOMES:
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h Day 6:predose
  Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)]; area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion [AUC(0-12), apparent terminal rate constant (λz), terminal half life (t1/2λz,h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration at steady state during dosing interval (Css,max), time to maximum concentration at steady state during dosing interval (tss,max), minimum plasma concentration at steady state during dosing interval (Css,min), area under the plasma concentration time curve from zero to time of the last quantifiable concentrations [AUC(0-t)], area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCτ); average plasma concentration during the dosing interval (Css,av), fluctuation index (FI, %)
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)]; area under the plasma concentration-time curve from zero to 8 hours after the start of the infusion [AUC(0-8), apparent terminal rate constant (λz), terminal half life (t1/2λz,h).
24 hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1,4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration at steady state during dosing interval (Css,max), time to maximum concentration at steady state during dosing interval (tss,max), minimum plasma concentration at steady state during dosing interval (Css,min), area under the plasma concentration time curve from zero to time of the last quantifiable concentrations [AUC(0-t)], area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCτ); average plasma concentration during the dosing interval (Css,av), fluctuation index (FI, %)
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1
  Amount of analyte excreted in the urine (Ae) during each interval and cumulatively, fraction of dose excreted into urine (fe,%) during each interval and cumulatively, total fraction of dose excreted in urine for all analytes combined (fe,total¬,%), and renal clearance (CLR).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 8
  Amount of analyte excreted in the urine (Ae,ss, mg) during each interval and cumulatively up to the end of the dosing interval, fraction of dose excreted into urine (fe,ss,%) during each interval and cumulatively up to the end of the dosing interval, total fraction of dose excreted in urine for all analytes combined (fe,ss,total ,%), and renal clearance (CLR,ss, L/h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)]; area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion [AUC(0-12), apparent terminal rate constant (λz), terminal half life (t1/2λz,h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration at steady state during dosing interval (Css,max), time to maximum concentration at steady state during dosing interval (tss,max), minimum plasma concentration at steady state during dosing interval (Css,min), area under the plasma concentration time curve from zero to time of the last quantifiable concentrations [AUC(0-t)], area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCτ); average plasma concentration during the dosing interval (Css,av), fluctuation index (FI, %)
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)]; area under the plasma concentration-time curve from zero to 8 hours after the start of the infusion [AUC(0-8), apparent terminal rate constant (λz), terminal half life (t1/2λz,h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration at steady state during dosing interval (Css,max), time to maximum concentration at steady state during dosing interval (tss,max), minimum plasma concentration at steady state during dosing interval (Css,min), area under the plasma concentration time curve from zero to time of the last quantifiable concentrations [AUC(0-t)], area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCτ); average plasma concentration during the dosing interval (Css,av), fluctuation index (FI, %)
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline M-1 following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)]; area under the plasma concentration-time curve from zero to 12 hours after the start of the infusion [AUC(0-12), apparent terminal rate constant (λz), terminal half life (t1/2λz,h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline M-1 following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration at steady state during dosing interval (Css,max), time to maximum concentration at steady state during dosing interval (tss,max), minimum plasma concentration at steady state during dosing interval (Css,min), area under the plasma concentration time curve from zero to time of the last quantifiable concentrations [AUC(0-t)], area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCτ); average plasma concentration during the dosing interval (Css,av), fluctuation index (FI,%)
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline M-1 following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration (Cmax), time to maximum concentration (tmax), area under the plasma concentration-time curve from zero to infinity (AUC), area under the plasma concentration-time curve from zero to time of the last quantifiable concentrations [AUC(0-t)]; area under the plasma concentration-time curve from zero to 8 hours after the start of the infusion [AUC(0-8), apparent terminal rate constant (λz), terminal half life (t1/2λz,h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline M-1 following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Maximum plasma concentration at steady state during dosing interval (Css,max), time to maximum concentration at steady state during dosing interval (tss,max), minimum plasma concentration at steady state during dosing interval (Css,min), area under the plasma concentration time curve from zero to time of the last quantifiable concentrations [AUC(0-t)], area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCτ); average plasma concentration during the dosing interval (Css,av), fluctuation index (FI, %)
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline fosamil following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1
  Amount of analyte excreted in the urine (Ae) during each interval and cumulatively, fraction of dose excreted into urine (fe,%) during each interval and cumulatively, total fraction of dose excreted in urine for all analytes combined (fe,total¬,%), and renal clearance (CL R).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline fosamil following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 8
  Amount of analyte excreted in the urine (Ae,ss, mg) during each interval and cumulatively up to the end of the dosing interval, fraction of dose excreted into urine (fe,ss,%) during each interval and cumulatively up to the end of the dosing interval, total fraction of dose excreted in urine for all analytes combined (fe,ss,total ,%), and renal clearance (CLR,ss, L/h).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline fosamil following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1
  Amount of analyte excreted in the urine (Ae) during each interval and cumulatively, fraction of dose excreted into urine (fe,%) during each interval and cumulatively, total fraction of dose excreted in urine for all analytes combined (fe,total¬,%), and renal clearance (CLR).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline fosamil following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 8
  Amount of analyte excreted in the urine (Ae,ss, mg) during each interval and cumulatively up to the end of the dosing interval, fraction of dose excreted into urine (fe,ss,%) during each interval and cumulatively up to the end of the dosing interval, total fraction of dose excreted in urine for all analytes combined (fe,ss,total ,%), and renal clearance (CLR,ss, L/h).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline M- 1 following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1
  Amount of analyte excreted in the urine (Ae) during each interval and cumulatively, fraction of dose excreted into urine (fe,%) during each interval and cumulatively, total fraction of dose excreted in urine for all analytes combined (fe,total¬,%), and renal clearance (CLR).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline M- 1 following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 8
  Amount of analyte excreted in the urine (Ae,ss, mg) during each interval and cumulatively up to the end of the dosing interval, fraction of dose excreted into urine (fe,ss,%) during each interval and cumulatively up to the end of the dosing interval, total fraction of dose excreted in urine for all analytes combined (fe,ss,total ,%), and renal clearance (CLR,ss, L/h).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline M- 1 following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1
  Amount of analyte excreted in the urine (Ae) during each interval and cumulatively, fraction of dose excreted into urine (fe,%) during each interval and cumulatively, total fraction of dose excreted in urine for all analytes combined (fe,total¬,%), and renal clearance (CLR).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline M- 1 following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 8
  Amount of analyte excreted in the urine (Ae,ss, mg) during each interval and cumulatively up to the end of the dosing interval, fraction of dose excreted into urine (fe,ss,%) during each interval and cumulatively up to the end of the dosing interval, total fraction of dose excreted in urine for all analytes combined (fe,ss,total ,%), and renal clearance (CLR,ss, L/h).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1
  Amount of analyte excreted in the urine (Ae) during each interval and cumulatively, fraction of dose excreted into urine (fe,%) during each interval and cumulatively, total fraction of dose excreted in urine for all analytes combined (fe,total¬,%), and renal clearance (CLR).
Urine pharmacokinetic parameters in terms of (see description) for ceftaroline following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 8
  amount of analyte excreted in the urine (Ae,ss, mg) during each interval and cumulatively up to the end of the dosing interval, fraction of dose excreted into urine (fe,ss,%) during each interval and cumulatively up to the end of the dosing interval, total fraction of dose excreted in urine for all analytes combined (fe,ss,total ,%), and renal clearance (CLR,ss, L/h).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h Day 6:predose
  Mean residence time (MRT), total body clearance of drug from plasma (CL for ceftaroline fosamil, apparent CL for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Apparent terminal rate constant (λz), terminal half-life (t½λz, h), accumulation ratio based on Cmax [Rac(Cmax)], accumulation ratio based on AUC [Rac(AUC)], and linearity factor.Mean residence time (MRT), plasma clearance at steady state (CLss for ceftaroline fosamil, apparent CLss for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Mean residence time (MRT), total body clearance of drug from plasma (CL for ceftaroline fosamil, apparent CL for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24 hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1,4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Apparent terminal rate constant (λz), terminal half-life (t½λz, h), accumulation ratio based on Cmax [Rac(Cmax)], accumulation ratio based on AUC [Rac(AUC)], and linearity factor. Mean residence time (MRT), plasma clearance at steady state (CLss for ceftaroline fosamil, apparent CLss for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following single dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Mean residence time (MRT), total body clearance of drug from plasma (CL for ceftaroline fosamil, apparent CL for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Apparent terminal rate constant (λz), terminal half-life (t½λz, h), accumulation ratio based on Cmax [Rac(Cmax)], accumulation ratio based on AUC [Rac(AUC)], and linearity factor.Mean residence time (MRT), plasma clearance at steady state (CLss for ceftaroline fosamil, apparent CLss for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following single dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Mean residence time (MRT), total body clearance of drug from plasma (CL for ceftaroline fosamil, apparent CL for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline fosamil following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Apparent terminal rate constant (λz), terminal half-life (t½λz, h), accumulation ratio based on Cmax [Rac(Cmax)], accumulation ratio based on AUC [Rac(AUC)], and linearity factor. Mean residence time (MRT), plasma clearance at steady state (CLss for ceftaroline fosamil, apparent CLss for ceftaroline), volume of distribution based on the terminal phase (Vz for ceftaroline fosamil, apparent Vz for ceftaroline), and volume of distribution at steady state (Vss for ceftaroline fosamil, apparent Vss for ceftaroline).
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline M-1 following multiple dose administration of ceftaroline fosamil 600 mg (every 12 h) 1 h infusion | Day 1, 4 and 8: Pre-dose, 20 min, 40 min, 55 min, 65 min, 75 min, 90 min, 120 min, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Apparent terminal rate constant (λz), terminal half-life (t½λz, h), accumulation ratio based on Cmax [Rac(Cmax)], accumulation ratio based on AUC [Rac(AUC)], and linearity factor.
24-hour plasma pharmacokinetic profile in terms of (see description) for ceftaroline M-1 following multiple dose administration of ceftaroline fosamil 600 mg (every 8 h) 2 h infusion | Day 1, 4 and 8: Pre-dose, 30 min, 60 min, 90 min, 115 min, 125 min, 2 h 15 min, 2.5 h, 3 h, 4 h, 6 h, 8 h, 12 h, 18 h 24 h,Day 6:predose
  Apparent terminal rate constant (λz), terminal half-life (t½λz, h), accumulation ratio based on Cmax [Rac(Cmax)], accumulation ratio based on AUC [Rac(AUC)], and linearity factor.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — AstraZeneca PharmaceuticalsC2C-7161800 Concord PikePO. Box 15437Wilmington De 19850-5437; Elizabeth Tranter, MBCHB MRCP, Principal Investigator — Hammersmith Medicines Cumberland Avenue London NW10 7EW UK; Mirjana Kujacic, MD, Study Chair — AstraZeneca Research and DevelopmentSE-431 83 MolndalSweden
Locations (1):
- Research site, London, United Kingdom

REFERENCES:
- [Derived] Das S, Li J, Iaconis J, Zhou D, Stone GG, Yan JL, Melnick D. Ceftaroline fosamil doses and breakpoints for Staphylococcus aureus in complicated skin and soft tissue infections. J Antimicrob Chemother. 2019 Feb 1;74(2):425-431. doi: 10.1093/jac/dky439. PMID 30380060
- [Derived] Yang L, Sunzel M, Xu P, Edeki T, Wilson D, Li J, Li H. Evaluation of the pharmacokinetics and safety of single and multiple ceftaroline fosamil infusions in healthy Chinese and Western subjects. Int J Clin Pharmacol Ther. 2015 Aug;53(8):681-91. doi: 10.5414/CP202343. PMID 26152131
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1376&filename=CSR-D3720C00010.pdf
- See also: CSR-D3720C00010.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1376&filename=CSR-D3720C00010.pdf
- See also: Clinical_Study_Protocol-Redacted-13.03.14 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1376&filename=D3720C00010_Clinical_Study_Protocol.pdf_Redacted-13.03.14.pdf